CLINICAL TRIAL: NCT01602913
Title: Incident Type II Diabetes Mellitus Among Patients Exposed to the Combination of Pravastatin and Paroxetine
Brief Title: Type II Diabetes Mellitus in Patients Exposed to Pravastatin and Paroxetine
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 116554; WEUSKOP5966 (Other: GSK)
Record Dates: First submitted 2012-05-10; First posted 2012-05-21 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Depression, Postpartum
Keywords: Pravastatin; Adverse Events; Type II Diabetes Mellitus; Incidence; Paroxetine
MeSH Terms: conditions — Depression, Postpartum; Diabetes Mellitus, Type 2 | interventions — Pravastatin; Paroxetine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with diagnosis of Type II Diabetes: Patients indicating T2DM after the index date (ICD-9-CM 250.x), or 1 diagnostic code and 1 prescription of oral anti-diabetic medications or insulin (or Byetta and Victoza) after the index date
  Interventions: Drug: Pravastatin alone; Drug: Paroxetine alone; Drug: Pravastatin and paroxetine combined
- Patients without diagnosis of Type II Diabetes: Patients not indicating T2DM
  Interventions: Drug: Pravastatin alone; Drug: Paroxetine alone; Drug: Pravastatin and paroxetine combined

INTERVENTIONS:
Drug: Pravastatin alone — Pravastatin is a member of the drug class of statins, also known as HMG-CoA reductase inhibitors, and is known to reduce the amount of cholesterol and other fatty substances in the blood. In addition, pravastatin is indicated to reduce the risk of myocardial infarction, revascularization and cardiovascular mortality in hypercholesterolemic patients who do not have clinically apparent coronary heart disease.
Drug: Paroxetine alone — Paroxetine is an orally administered selective serotonin reuptake inhibitor (SSRI) for the treatment of depression
Drug: Pravastatin and paroxetine combined — Pravastatin is a member of the drug class of statins, also known as HMG-CoA reductase inhibitors, and is known to reduce the amount of cholesterol and other fatty substances in the blood. In addition, pravastatin is indicated to reduce the risk of myocardial infarction, revascularization and cardiovascular mortality in hypercholesterolemic patients who do not have clinically apparent coronary heart disease. Paroxetine is an orally administered selective serotonin reuptake inhibitor (SSRI) for the treatment of depression

SUMMARY:
Type 2 Diabetes (T2DM) is a life-long, chronic condition affecting an individuals' ability to regulate glucose levels in the blood. Diabetes can cause many severe complications if not treated properly. Hyperglycemia is a regular effect of uncontrolled diabetes and can lead to complications such as cardiovascular disease, chronic renal failure, diabetic retinopathy and inability to maintain a healthy body weight.

Cardiovascular Disease (CVD) is now the leading cause of death worldwide, affecting millions of people in both developed and non-developed countries. The buildup of cholesterol in the bloodstream may cause the excess to be deposited in the coronary arteries of the heart and the carotid arteries of the brain. The cholesterol deposits are a factor of the plaques that cause blockage of the arteries which can in turn lead to heart disease and stroke. By lowering the blood levels of cholesterol, risks of heart disease, strokes and heart attacks are reduced. Medications such as HMG-CoA reductase inhibitors and fibrates are useful in the prevention of CVD.

Pravastatin is a member of the drug class of statins, also known as HMG-CoA reductase inhibitors, and is shown as an adjunctive therapy to diet. It is known to reduce the amount of cholesterol and other fatty substances in the blood. In addition, pravastatin is indicated to reduce the risk of myocardial infarction, revascularization and cardiovascular mortality in hypercholesterolemic patients who do not have clinically apparent coronary heart disease. The recommended starting dose for adults is 40 mg once daily. For patients who do not reach the LDL-C goal with 40 mg, it is recommended to use an 80 mg dose. For persons with significant renal impairment the recommended dose is 10 mg. Children aged 8-13 years have a recommended starting dose of 20 mg daily. Adolescents aged 14 to 18 years have a recommended starting dose of 40 mg daily.

Depression is known as the most common mental disorder and most prevalent type of mood disorder today. It can be seen as a state of mood, a symptom, a syndrome or as a clinical diagnosis. Depression is a common disorder, affecting about 121 million people worldwide. Depression is more likely to co-occur with medical illnesses such as stroke, heart disease, cancer and diabetes. Up to one-quarter of people with diabetes are estimated to experience depression which is two times more than those who do not suffer from diabetes. Studies have shown that major depression mainly occurs in 2¬4 percent of people in the community, in 5-10 percent of primary care patients and 10-14 percent of medical inpatients. Also, recent studies have estimated that the symptoms continue over a 6 month to one year period in patients with major depression. The severity of the symptoms and the incidence of medical illness are expected to predict the persistence of depression. Depression can be treated effectively by a variety of antidepressants and/or psychotherapies. If treated appropriately, over 80 percent of people who suffer from depression can be helped.

Paroxetine is an orally administered selective serotonin reuptake inhibitor (SSRI) antidepressant. It was the first antidepressant that was formally approved in the United States for the treatment of panic attacks, major depression, post¬traumatic stress disorder, social anxiety, generalized anxiety disorder, panic disorder and obsessive-compulsive disorder. Paroxetine has a well-established safety profile and it shares the common side effects and contraindications of other SSRI's which include nausea and somnolence and is associated with weight gain.

This study proposes to conduct a retrospective cohort study to assess the risk of new onset diabetes among patients undergoing treatment with Pravastatin or other statins, and Paroxetine or other SSRI's. This study will compare the risk of co administration of two drug classes versus the use of each agent alone. In addition, the risk among patients prescribed Paroxetine and fibrates in combination, relative to the use of Paroxetine singly, will be examined to determine whether any interaction found between Paroxetine and statins extends to other drugs indicated for hypercholesterolemia.

The first primary objective of the study is to estimate the incidence of Type 2 Diabetes (T2DM) among patients newly exposed to pravastatin in combination with paroxetine, or other SSRIs, compared to those newly exposed to pravastatin alone. The second primary objective is to estimate the incidence of Type 2 Diabetes (T2DM) among patients newly exposed to paroxetine in combination with pravastatin, other statins, or fibrates, compared to those newly exposed to paroxetine alone.

ELIGIBILITY:
Inclusion Criteria:

* patients 18 years of age or older at the index date
* patients newly prescribed pravastatin or paroxetine
* patients enrolled in the database for at least 180 days prior to the index date

Exclusion Criteria:

* patients prescribed any statins, fibrates, or SRRIs other than the one defined per cohort during the duration of follow-up (in- class medication switching will result in censoring at the date of switch);
* patients with T2DM or gestational diabetes ever recorded in their record
* patients with impaired glucose tolerance ever recorded in their record
* patients ever prescribed any oral anti-diabetic medications or insulin; or injectable GLP¬1 analogues
* patients considered to have Type 1 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data will be ascertained from the Thomson-Reuters Marketscan database, which contains administrative healthcare data among an insured population in the US between 2000 and 2009. The MarketScan® Databases capture person-specific clinical utilization, expenditures, and enrollment across inpatient, outpatient, and prescription drug from a selection of large employers, health plans, and government and public organizations (MarketScan Users manual). The MarketScan Databases link paid claims and encounter data to detailed patient information across sites and types of providers, and over time. The annual medical databases include private sector health data from approximately 100 payers. Historically, more than 500 million claim records are available in the MarketScan Databases. These data represent the medical experience of insured employees and their dependents for active employees, early retirees, COBRA continues and Medicare-eligible retirees with employer-provided Medicare supplemental
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-12; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Incidence of T2DM defined as having at least 2 diagnostic codes indicating T2DM after the index date, or 1 diagnostic code and 1 prescription of oral anti-diabetic medications or insulin (or Byetta and Victoza) after the index date | Up to ten years

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline